CLINICAL TRIAL: NCT00605137
Title: Safety of Insulin Detemir and Insulin NPH in Children With Type 1 Diabetes Mellitus
Brief Title: Safety of Insulin Detemir in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1604; JapicCTI-R070014 (Registry Identifier: japic)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin NPH

SUMMARY:
This trial is conducted in Japan. The aim of trial is to investigate the safety of insulin detemir and insulin NPH in children with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least one year
* Current treatment of basal-bolus regimen for at least 12 weeks using an intermediate/long-acting human insulin and insulin aspart and/or soluble human insulin
* HbA1C below 11.0%
* Willing to comply with Investigator's instructions
* Able and willing to perform self-monitoring of capillary blood glucose and to take measures in case of hypoglycaemia

Exclusion Criteria:

* Impaired renal function
* Impaired hepatic function
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia (as judged by the Investigator or Sub-Investigator)
* Proliferative retinopathy or maculopathy requiring acute treatment
* Uncontrolled treated/untreated hypertension
* Current treatment with total daily insulin dose of more than 2.00 IU/kg
* Current treatment or expected at the screening to start treatment with systemic corticosteroids

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2004-05-21 (Actual); Primary Completion 2005-04-23 (Actual); Study Completion 2005-04-23 (Actual)

PRIMARY OUTCOMES:
Incidence of hypoglycaemic episodes | during treatment

SECONDARY OUTCOMES:
Adverse events
Laboratory assessments and other safety endpoints
HbA1C, self monitored blood glucose and within-subject variability of glucose
Height
Insulin doses

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com